CLINICAL TRIAL: NCT05605314
Title: Clinical Cohort Study in Patients With Different Subtypes of Primary Sjogren Syndrome Related Dry Eye
Acronym: pSS
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: fengyun77470
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pSS-DED: DED patients who visited the dry eye clinic of Peking University Third Hospital from 2021 to May 2028. The pSS-DED patients further accepted the diagnosis of rheumatology department. All enrolled DED participants met the criterion of TFOS DEWS II Definition and Classification Report and pSS-DED group also met 2016ACR/EULAR pSS diagnosis and classification consensus.
  Interventions: Other: Cyclosporine
- nss-DED: DED patients who visited the dry eye clinic of Peking University Third Hospital from 2021 to May 2028.
  Interventions: Other: Cyclosporine

INTERVENTIONS:
Other: Cyclosporine — eye drop

SUMMARY:
Primary Sjögren's syndrome is a chronic autoimmune disease that primarily involves exocrine glands, most commonly manifested in dry eye, dry mouth, and in other systems of the body.

DETAILED DESCRIPTION:
Patients usually first seek for the ophthalmologist for severe dry eye symptoms, and most clinicians are ill-informed about Sjögren's syndrome dry eye disease (SS-DED), which can lead to missed diagnoses and misdiagnoses. Clinically, there are not many types of patients with pSS and the number of in-depth studies is small. Meanwhile, there are no specific drugs for the treatment of SS-DED, and most patients need to be treated with multiple methods to understand which methods are most effective. In this study, by establishing a clinical cohort of patients with different subtypes of dry eye with pSS, we explored the association between the primary organs affected by pSS and various biomarkers related to tear fluid and blood, and the association between the primary organs affected by pSS, tear components and blood markers and the severity of ocular involvement, symptom progression and prognosis. This study initially constructs a special cohort of patients with pSS ocular involvement, which may explain its pathogenesis from a new perspective in diagnose, classification and treatment.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled DED participants met the criterion of TFOS DEWS II Definition and Classification Report and pSS-DED group also met 2016ACR/EULAR pSS diagnosis and classification consensus.

Exclusion Criteria:

* (1) patients were diagnosed as any rheumatic or systematic diseases that would probably affect tear function except for pSS and DED. (2) had a history of ocular trauma or surgery. (3) had a history of wearing contact lens. (4) had concomitant ocular lesions such as acute inflammation or infection, glaucoma or eyelid abnormalities. (5) cannot cooperate properly or finish related examinations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pSS and DED patients who visited the dry eye clinic of Peking University Third Hospital from January 2021 to January 2028.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
ESSDAI | 2021.1~2028.1
  Fill out the scale

SECONDARY OUTCOMES:
Schirmer | 2021.1~2028.1
  The Schirmer I test was performed without topical anesthesia after all other examinations by slit lamp had been completed at least 15 minutes to avoid any effect of keratoconjunctival staining. A Schirmer test strip (Liaoning Meizilin Pharmaceutical Co., Ltd.) was placed on the outer one third of the temporal lower conjunctival fornix for 5 min. The strip was then removed, and the length of the wet filter paper was recorded in millimeters.
BUT，TMH | 2021.1~2028.1
  All participants were instilled a minimal volume fluorescein into the inferior temporal tear meniscus by fluorescein sodium ophthalmic test paper (Liaoning Meizilin Pharmaceutical Co., Ltd.) for the evaluation of tear menicus height (TMH) and fluorescein tear break-up time (FBUT) during slit lamp examination. Then, patients were asked to blink several times to ensure adequate mixing of the fluorescein dye with the tears. Under the cobalt blue light of the slit lamp microscope, TMH were recorded and the time interval between the last complete blink and the appearance of the first corneal dark spot was timed using a stopwatch. The average of three measurements was recorded as the FBUT.

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Tao, PhD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No